CLINICAL TRIAL: NCT00711750
Title: Immediate Maintained Cannulation of a Newly Implanted Prosthetic Arteriovenous Access for Acute Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: FEMH-96042
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: End-Stage Renal Disease; Prosthetic Arteriovenous Access
Keywords: underwent; specific; creation; hospital; November 2003; October 2005
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Objectives: Examine the acute utility of immediate maintained cannulations of a newly implanted prosthetic arteriovenous access. Background: Recurrent failure of central catheterization is not uncommon. An alternative access is necessary for acute hemodialysis after the exhaustion of central veins. Methods: We constructed the access by cannulating two dialysis needle-catheters and securing them on the skin after the implantation of the graft. The access was used immediately and maintained for one week and thereafter used as a long-term access.

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease underwent the specific prosthetic arteriovenous access creation in our hospital from November 2003 to October 2005

Exclusion Criteria:

* patients' poor health as long as they did not have other options and needed an access for acute hemodialysis. Exclusions included shock, active systemic infection, and rejection by the attending nephrologists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end-stage renal disease underwent the specific prosthetic arteriovenous access creation in our hospital from November 2003 to October 2005 were retrospectively reviewed.
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan